CLINICAL TRIAL: NCT02059096
Title: Analgesic Effect of Repetitive Transcranial Magnetic Stimulation (rTMS) for Central Neuropathic Pain in Multiple Sclerosis
Acronym: STIMASEP
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHU-0179; 2013-A01422-43
Record Dates: First submitted 2014-02-06; First posted 2014-02-11 (Estimated); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Multiple Sclerosis With Central Neuropathic Pain
Keywords: Multiple Sclerosis; Repetitive transcranial magnetic stimulation (rTMS); Chronic neuropathic pain; Cortical excitability
MeSH Terms: conditions — Multiple Sclerosis | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Repetitive transcranial magnetic stimulation (rTMS) (Experimental): The goal of this study is to compare the analgesic effects of two types of primary Motor cortex (M1) rTMS, namely 10Hz and prolonged continuous Theta-Burst Stimulation (pcTBS), with sham stimulation
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)
- Theta-Burst Stimulation (pcTBS) (Other): The goal of this study is to compare the analgesic effects of two types of primary Motor cortex (M1) rTMS, namely 10Hz and prolonged continuous Theta-Burst Stimulation (pcTBS), with sham stimulation.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)
- repetitive Transcranial Magnetic Stimulation (rTMS)placebo (Other): The goal of this study is to compare the analgesic effects of two types of primary Motor cortex (M1) rTMS, namely 10Hz and prolonged continuous Theta-Burst Stimulation (pcTBS), with sham stimulation.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (rTMS)

SUMMARY:
This study is designed to evaluate the effect of repetitive Transcranial Magnetic Stimulation (rTMS) in the resolution of chronic pain. Participants will be patients with Multiple Sclerosis suffering from chronic pain of neurological origin.

DETAILED DESCRIPTION:
On the one hand, Multiple Sclerosis (MS) is the most frequent chronic disease generating neurological disability in young adults. Among the many types of disabilities associated with MS, chronic pain is very frequent, especially neuropathic pain. This type of pain is often treatment resistant. Moreover, abnormal intra-cortical excitability has been described in MS patients.

On the other hand, repetitive Transcranial Magnetic Stimulation (rTMS) has shown an analgesic effect in various chronic pain conditions (fibromyalgia, post-stroke, peripheral neuropathic pain). Three groups have shown that analgesia was correlated to defective intra-cortical excitability restoration.

The goal of this study is to compare the analgesic effects of two types of primary Motor cortex (M1) rTMS, namely 10Hz and prolonged continuous Theta-Burst Stimulation (pcTBS), with sham stimulation.

Patients will benefit from 1 daily session per day for 5 consecutive days and from a total follow up of 4 weeks. Pain will be assessed each day and several other signs and symptoms will be repeatedly assessed.

ELIGIBILITY:
Inclusion Criteria:

* relapsing-remitting Multiple Sclerosis
* 18 to 60 years
* central neuropathic pain with a DN4 score of 4 or more out of 10
* average pain of at least 4/10
* presence of pain at least 4 days per week
* presence of pain for at least 3 months
* stable analgesic treatment

Exclusion Criteria:

* relapse during the previous 30 days
* contraindication for rTMS
* peripheral neuropathic pain
* severe depression
* epilepsia
* resting motor threshold above 75%

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2014-01-05 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in "average pain" score on the brief pain inventory | at day 8
  Variation of the "Average pain" score on the Brief Pain Inventory between before treatment (on a 7 days period) and day 8.

SECONDARY OUTCOMES:
change from baseline in "average pain" score on the brief pain inventory | at weekk 3 and 4
  Variation of the average pain at several time-points during the 4 weeks follow-up
Location of MRI abnormalities | at week 3 and 4
  Correlation between pain and pain decrease with MRI abnormalities in several regions of interest
Intra-cortical excitability evaluated by motor threshold, MEP amplitude, SICI and ICF | at week 3 and 4
Number of participants with adverse events as a measure of safety and tolerability | at day 1
change from baseline in specific questionnaires | at day 8, week 3 and 4

CONTACTS AND LOCATIONS:
Overall Officials: Xavier MOISSET, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (3):
- France (3):
  - CHU Ambroise Paré, Boulogne-Billancourt
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - Hôpital Henri Mondor, Créteil